CLINICAL TRIAL: NCT04801901
Title: PRESERVE Radial: A PRospEctive Randomized Clinical Study Comparing Radial ArtERy Intimal Hyperplasia Following Distal Vs. ForEarm TransRadial Arterial Access for Coronary Angiography
Brief Title: Distal Transradial Access for Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Wayne B. Batchelor M.D., Director of Interventional Cardiology, Inova Heart and Vascular Institute, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U20-04-4021
Record Dates: First submitted 2021-01-07; First posted 2021-03-17 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Transradial Access; Coronary Angiography; Radial Artery Intimal Medial Thickness; Distal Radial Artery Access (dTRA)

STUDY DESIGN:
Intervention Model Description: Prospective randomized non-blinded study evaluating whether distal radial artery access (dTRA) from the anatomic snuffbox is associated with less trauma and adverse remodeling to the forearm radial artery compared to standardard forearm radial access (fTRA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal transradial access (dTRA) (Experimental): Subjects randomized to the experimental arm will undergo left heart catheterization using distal transradial access (dTRA) to facilitate coronary angiography and/or percutaneous coronary intervention.
  Interventions: Procedure: dTRA
- Forearm radial access (fTRA) (Active Comparator): Cardiac catheterization to facilitate coronary angiography and/or percutaneous coronary intervention using the standard forearm radial artery which is the current standard of care in interventional cardiology.
  Interventions: Procedure: fTRA

INTERVENTIONS:
Procedure: dTRA — Subjects randomized to the experimental arm will undergo left heart catheterization, coronary angiography and/or percutaneous coronary intervention using distal transradial access (dTRA)
  Arms: Distal transradial access (dTRA)
Procedure: fTRA — Left heart catheterization, coronary angiography and/or percutaneous coronary intervention using the left forearm radial artery.
  Arms: Forearm radial access (fTRA)

SUMMARY:
Prospective randomized non-blinded study to determine degree of vessel trauma and adverse remodeling of the proximal forearm radial artery following distal radial artery access (dTRA) for cardiac catheterization compared to standard forearm transradial access (fTRA).

DETAILED DESCRIPTION:
To determine degree of vessel trauma and adverse remodeling of the proximal forearm radial artery, using ultrahigh resolution (55 MHz) ultrasound, following distal radial artery access (dTRA) for cardiac catheterization compared to standard forearm transradial access (fTRA) at 90 days post-procedure. Secondary outcome measures will include metrics of procedural success at 24 hours, as well as functional assessment of pain and motor strength of the ipsilateral upper extremity at 90 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients undergoing elective and non-emergent TR LHC and/or PCI at the INOVA Heart and Vascular Institute
2. Able to provide informed consent.
3. Patients willing to complete a 90day post PCI radial artery ultrasound.

Exclusion Criteria:

1. Patients with previous cannulation of both the right and left forearm RA's for coronary angiography and/or PCI. In patients with prior cannulation of one RA, the contralateral arm may be used for this study.
2. Patients who are not willing to undergo the necessary follow-up ultrasound examinations.
3. ST elevation myocardial infarction or other emergent PCI
4. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Radial artery intimal medial thickness following dTRA and fTRA | 90 days post-cardiac catheterization.
  Intimal medial thickness (mm) of the forearm radial artery followed dTRA and fTRA as assessed using ultrahigh resolution 55 MHz ultrasound probe at 90 days post cardiac catheterization.

SECONDARY OUTCOMES:
Radial artery trauma followed dTRA and fTRA | 90 days post-cardiac catheterization
  Number of participants with limited access site intimal tears, dissections, thrombosis, occlusions and pseudoaneurysms of the radial artery as assessed using ultrahigh resolution 55 MHz ultrasound at the site of puncture at 90 days post cardiac catheterization
Functional assessment of the ipsilateral upper extremity following dTRA and fTRA | 90 days post-cardiac catheterization
  Pain and motor strength of the ipsilateral upper extremity using the Borg (0-none to 10-maximal) and Disabilities of the Arm, Shoulders and Hand (DASH) (0-no disability to 100-most severe disability) scales 90 days post-cardiac catheterization.
Number of cannulation attempts | 24 hours post-cardiac catheterization
  Number of cannulation attempts prior to achieving successful vascular access
Radial artery access time | 24 hours post-cardiac catheterization
  Time (minutes) from initial attempt to successful access of the radial artery.
Access site crossover | 24 hours post-cardiac catheterization
  Number of patients with failure of radial artery cannulation requiring crossover to alternative radial artery access or transfemoral access
Total procedural time | 24 hours post-cardiac catheterization
  Total procedural time (minutes) from time of access to completion of the cardiac catheterization.
Duration of hemostasis | 24 hours post-cardiac catheterization
  Total duration of hemostasis (minutes) following completion of cardiac catheterization
Incidence of hematomas | 24 hours post-cardiac catheterization
  Number of patients with EASY Class III or greater hematomas
Percutaneous Coronary Intervention Success | 24 hours post-cardiac catheterization
  Achievement of Thrombolysis in Myocardial Infarction (TIMI) 3 flow following percutaneous coronary intervention
Coronary dissection | 24 hours post-cardiac catheterization
  Iatrogenic coronary dissection at the of cardiac catheterization
Myocardial infarction requiring revascularization | 24 hours post-cardiac catheterization
  Periprocedural myocardial infarction requiring urgent revascularization within 24 hours post-cardiac catheterization.

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data including demographics, cardiac history indications for cardiac catheterization and all follow up data related to primary outcome, secondary ultrasound endpoints, interventional endpoints and secondary functional outcomes will be shared.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Campeau L. Percutaneous radial artery approach for coronary angiography. Cathet Cardiovasc Diagn. 1989 Jan;16(1):3-7. doi: 10.1002/ccd.1810160103. PMID 2912567
- [Background] Ferrante G, Rao SV, Juni P, Da Costa BR, Reimers B, Condorelli G, Anzuini A, Jolly SS, Bertrand OF, Krucoff MW, Windecker S, Valgimigli M. Radial Versus Femoral Access for Coronary Interventions Across the Entire Spectrum of Patients With Coronary Artery Disease: A Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2016 Jul 25;9(14):1419-34. doi: 10.1016/j.jcin.2016.04.014. Epub 2016 Jun 29. PMID 27372195
- [Background] Kopin D, Seth M, Sukul D, Dixon S, Aronow HD, Lee D, Tucciarone M, Pielsticker E, Gurm HS. Primary and Secondary Vascular Access Site Complications Associated With Percutaneous Coronary Intervention: Insights From the BMC2 Registry. JACC Cardiovasc Interv. 2019 Nov 25;12(22):2247-2256. doi: 10.1016/j.jcin.2019.05.051. Epub 2019 Aug 28. PMID 31473240
- [Background] Valle JA, Kaltenbach LA, Bradley SM, Yeh RW, Rao SV, Gurm HS, Armstrong EJ, Messenger JC, Waldo SW. Variation in the Adoption of Transradial Access for ST-Segment Elevation Myocardial Infarction: Insights From the NCDR CathPCI Registry. JACC Cardiovasc Interv. 2017 Nov 27;10(22):2242-2254. doi: 10.1016/j.jcin.2017.07.020. Epub 2017 Nov 1. PMID 29102582
- [Background] Mason PJ, Shah B, Tamis-Holland JE, Bittl JA, Cohen MG, Safirstein J, Drachman DE, Valle JA, Rhodes D, Gilchrist IC; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; and Council on Genomic and Precision Medicine. An Update on Radial Artery Access and Best Practices for Transradial Coronary Angiography and Intervention in Acute Coronary Syndrome: A Scientific Statement From the American Heart Association. Circ Cardiovasc Interv. 2018 Sep;11(9):e000035. doi: 10.1161/HCV.0000000000000035. PMID 30354598
- [Background] Rashid M, Kwok CS, Pancholy S, Chugh S, Kedev SA, Bernat I, Ratib K, Large A, Fraser D, Nolan J, Mamas MA. Radial Artery Occlusion After Transradial Interventions: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Jan 25;5(1):e002686. doi: 10.1161/JAHA.115.002686. PMID 26811162
- [Background] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Background] Babunashvili A, Dundua D. Recanalization and reuse of early occluded radial artery within 6 days after previous transradial diagnostic procedure. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):530-6. doi: 10.1002/ccd.22846. PMID 20939038
- [Background] Aoi S, Htun WW, Freeo S, Lee S, Kyaw H, Alfaro V, Coppola J, Pancholy S, Kwan T. Distal transradial artery access in the anatomical snuffbox for coronary angiography as an alternative access site for faster hemostasis. Catheter Cardiovasc Interv. 2019 Nov 1;94(5):651-657. doi: 10.1002/ccd.28155. Epub 2019 Feb 24. PMID 30801939
- [Background] Koutouzis M, Kontopodis E, Tassopoulos A, Tsiafoutis I, Katsanou K, Rigatou A, Didagelos M, Andreou K, Lazaris E, Oikonomidis N, Maniotis C, Ziakas A. Distal Versus Traditional Radial Approach for Coronary Angiography. Cardiovasc Revasc Med. 2019 Aug;20(8):678-680. doi: 10.1016/j.carrev.2018.09.018. Epub 2018 Oct 2. PMID 30314833
- [Background] Nairoukh Z, Jahangir S, Adjepong D, Malik BH. Distal Radial Artery Access: The Future of Cardiovascular Intervention. Cureus. 2020 Mar 7;12(3):e7201. doi: 10.7759/cureus.7201. PMID 32269880
- [Background] Shroff AR, Gulati R, Drachman DE, Feldman DN, Gilchrist IC, Kaul P, Lata K, Pancholy SB, Panetta CJ, Seto AH, Speiser B, Steinberg DH, Vidovich MI, Woody WW, Rao SV. SCAI expert consensus statement update on best practices for transradial angiography and intervention. Catheter Cardiovasc Interv. 2020 Feb;95(2):245-252. doi: 10.1002/ccd.28672. Epub 2019 Dec 27. PMID 31880380
- [Background] Roghani-Dehkordi F, Hashemifard O, Sadeghi M, Mansouri R, Akbarzadeh M, Dehghani A, Akbari M. Distal accesses in the hand (two novel techniques) for percutaneous coronary angiography and intervention. ARYA Atheroscler. 2018 Mar;14(2):95-100. doi: 10.22122/arya.v14i2.1743. PMID 30108641
- [Background] Sgueglia GA, Di Giorgio A, Gaspardone A, Babunashvili A. Anatomic Basis and Physiological Rationale of Distal Radial Artery Access for Percutaneous Coronary and Endovascular Procedures. JACC Cardiovasc Interv. 2018 Oct 22;11(20):2113-2119. doi: 10.1016/j.jcin.2018.04.045. PMID 30336816
- [Background] Batchelor W, Dahya V, McGee D, Katopodis J, Dixon W, Campbell J, Meredith A, Knap P, Parkin M, Noel T. Ultrahigh-resolution ultrasound characterization of access site trauma and intimal hyperplasia following use of a 7F sheathless guide versus 6F sheath/guide combination for transradial artery PCI: Results of the PRAGMATIC trial. Am Heart J. 2018 Apr;198:75-83. doi: 10.1016/j.ahj.2017.11.017. Epub 2017 Dec 15. PMID 29653651
- [Background] Sarkola T, Slorach C, Hui W, Bradley TJ, Redington AN, Jaeggi E. Transcutaneous very-high resolution ultrasound for the quantification of carotid arterial intima-media thickness in children - feasibility and comparison with conventional high resolution vascular ultrasound imaging. Atherosclerosis. 2012 Sep;224(1):102-7. doi: 10.1016/j.atherosclerosis.2012.06.054. Epub 2012 Jun 27. PMID 22784638
- [Background] Stegemann E, Sansone R, Stegemann B, Kelm M, Heiss C. Validation of High-Resolution Ultrasound Measurements of Intima-Media Thickness of the Radial Artery for the Assessment of Structural Remodeling. Angiology. 2015 Jul;66(6):574-7. doi: 10.1177/0003319714544699. Epub 2014 Aug 5. PMID 25100749
- [Background] Costa F, van Leeuwen MA, Daemen J, Diletti R, Kauer F, van Geuns RJ, Ligthart J, Witberg K, Zijlstra F, Valgimigli M, Van Mieghem NM. The Rotterdam Radial Access Research: Ultrasound-Based Radial Artery Evaluation for Diagnostic and Therapeutic Coronary Procedures. Circ Cardiovasc Interv. 2016 Feb;9(2):e003129. doi: 10.1161/CIRCINTERVENTIONS.115.003129. PMID 26839392
- [Background] Foster FS, Mehi J, Lukacs M, Hirson D, White C, Chaggares C, Needles A. A new 15-50 MHz array-based micro-ultrasound scanner for preclinical imaging. Ultrasound Med Biol. 2009 Oct;35(10):1700-8. doi: 10.1016/j.ultrasmedbio.2009.04.012. Epub 2009 Aug 3. PMID 19647922
- [Background] Jester A, Harth A, Wind G, Germann G, Sauerbier M. Disabilities of the arm, shoulder and hand (DASH) questionnaire: Determining functional activity profiles in patients with upper extremity disorders. J Hand Surg Br. 2005 Feb;30(1):23-8. doi: 10.1016/j.jhsb.2004.08.008. PMID 15620487
- [Background] Shroff A, Siddiqui S, Burg A, Singla I. Identification and management of complications of transradial procedures. Curr Cardiol Rep. 2013 Apr;15(4):350. doi: 10.1007/s11886-013-0350-x. PMID 23420446
- [Background] Pancholy S, Coppola J, Patel T, Roke-Thomas M. Prevention of radial artery occlusion-patent hemostasis evaluation trial (PROPHET study): a randomized comparison of traditional versus patency documented hemostasis after transradial catheterization. Catheter Cardiovasc Interv. 2008 Sep 1;72(3):335-340. doi: 10.1002/ccd.21639. PMID 18726956
- [Derived] Tehrani BN, Sherwood MW, Damluji AA, Epps KC, Bakhshi H, Cilia L, Dassanayake I, Eltebaney M, Gattani R, Howard E, Kepplinger D, Ofosu-Somuah A, Batchelor WB. A Randomized Comparison of Radial Artery Intimal Hyperplasia Following Distal Versus Proximal Transradial Access for Coronary Angiography: PRESERVE RADIAL. J Am Heart Assoc. 2024 Feb 20;13(4):e031504. doi: 10.1161/JAHA.123.031504. Epub 2024 Feb 14. PMID 38353242